CLINICAL TRIAL: NCT00335894
Title: A Prospective, Randomized, Investigator-blind, Controlled, Clinical Study of Phase III on the Efficacy and Tolerability of hMG-IBSA (IBSA) vs Menopur (Ferring) Administered s.c. in Women Undergoing COH in an ART Programme (IVF)
Brief Title: Clinical Study of Clinical Efficacy and Tolerability of hMG-IBSA s.c.in Women Undergoing COH in an ART Programme (IVF).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04I/HMG10
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2008-12

CONDITIONS: Infertility
Keywords: Infertility; IVF; ART; hMG
MeSH Terms: conditions — Infertility | interventions — hMG-IBSA

INTERVENTIONS:
Drug: hMG-IBSA

SUMMARY:
Multicenter, prospective, randomized, investigator blind, controlled clinical trial. Two parallel groups, one receiving the test drug hMG (hMG-IBSA, IBSA Institut Biochimique sa) and the other the reference drug hMG (Menopur, Ferring Pharmaceuticals, Inc.).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the clinical efficacy and general tolerability of two different subcutaneous hMG preparations (hMG-IBSA, IBSA vs Menopur, Ferring Pharmaceuticals, Inc.) when administered to patients undergoing controlled ovarian stimulation for IVF.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing ovarian stimulation for IVF with or without ICSI (intracytoplasmic sperm injection) and with the following characteristics:
* Voluntary given informed consent to study participation in writing encompassing consent to data recording and verification procedures;
* > 18/= and < 37 years old;
* BMI between 18 and 28 kg/m2;
* Less than 3 previous completed IVF cycles;
* Basal FSH level less than 10 IU/L once within 6 months prior to the study;
* Within 12 month of the beginning of the study, uterine cavity consistent with expected normal function as assessed through a hysterosalpingogram, or sonohysterogram, or hysteroscopic examination or TVUS;
* Normal or clinically insignificant haematology and blood chemistry values.

Exclusion Criteria:

* Primary ovarian failure or women known as poor responders;
* Signs of PCO, according to the Rotterdam Criteria;
* At least one ovary inaccessible for oocyte retrieval;
* One or more ovarian cysts > 10 mm;
* Hydrosalpinx that have not been surgically removed or ligated;
* Stage III or IV endometriosis;
* Patients affected by pathologies associated with any contraindication of being pregnant;
* Hypersensitivity to the study medication;
* Abnormal bleeding of undetermined origin;
* Uncontrolled thyroid or adrenal dysfunction;
* Neoplasias;
* PAP smear III within the last 2 years;
* Severe impairment of the renal and/or hepatic functions;
* Lactation;
* Hyperprolactinaemia;
* Participation in a concurrent clinical trial or in another trial within the past four weeks;
* Use of concomitant medication that might interfere with study evaluations.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2009-03

PRIMARY OUTCOMES:
total number of oocytes retrieved 34 - 36 hours after hCG administration.

SECONDARY OUTCOMES:
Total dose of hMG (IU); number of days of hMG stimulation and stimulation duration; cancellation rate with reasons; 17β-estradiol (E2) serum concentration; number of follicles >16 mm.
number of mature oocytes and inseminated oocytes; fertilization rate.
embryo score; number of transferred embryos; implantation rate, number of transferred embryos; clinical pregnancy rate
Tolerability evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Placido, Prof, Study Director — Federico II University
Locations (2):
- Italy (2):
  - Università degli Studi di Bologna, Bologna, Bologna
  - Università degli Studi di Napoli Federico II, Napoli, Napoli

REFERENCES:
- [Background] Hauschke D, Kieser M, Diletti E, Burke M. Sample size determination for proving equivalence based on the ratio of two means for normally distributed data. Stat Med. 1999 Jan 15;18(1):93-105. doi: 10.1002/(sici)1097-0258(19990115)18:13.0.co;2-8. PMID 9990695
- [Background] Veeck LL. Oocyte assessment and biological performance. Ann N Y Acad Sci. 1988;541:259-74. doi: 10.1111/j.1749-6632.1988.tb22263.x. No abstract available. PMID 3195909
- [Background] GEMZELL CA, DICZFALUSY E, TILLINGER G. Clinical effect of human pituitary follicle-stimulating hormone (FSH). J Clin Endocrinol Metab. 1958 Dec;18(12):1333-48. doi: 10.1210/jcem-18-12-1333. No abstract available. PMID 13611018
- [Background] Filicori M, Cognigni GE, Pocognoli P, Tabarelli C, Ferlini F, Perri T, Parmegiani L. Comparison of controlled ovarian stimulation with human menopausal gonadotropin or recombinant follicle-stimulating hormone. Fertil Steril. 2003 Aug;80(2):390-7. doi: 10.1016/s0015-0282(03)00594-6. PMID 12909504
- [Background] Kilani Z, Dakkak A, Ghunaim S, Cognigni GE, Tabarelli C, Parmegiani L, Filicori M. A prospective, randomized, controlled trial comparing highly purified hMG with recombinant FSH in women undergoing ICSI: ovarian response and clinical outcomes. Hum Reprod. 2003 Jun;18(6):1194-9. doi: 10.1093/humrep/deg252. PMID 12773445
- [Background] Thompson CR, Hansen LM. Pergonal (menotropins): a summary of clinical experience in the induction of ovulation and pregnancy. Fertil Steril. 1970 Dec;21(12):844-53. doi: 10.1016/s0015-0282(16)37925-0. No abstract available. PMID 5481991
- [Background] Oelsner G, Serr DM, Mashiach S, Blankstein J, Snyder M, Lunenfeld B. The study of induction of ovulation with menotropins: analysis of results of 1897 treatment cycles. Fertil Steril. 1978 Nov;30(5):538-44. doi: 10.1016/s0015-0282(16)43634-4. No abstract available. PMID 720642
- [Background] Schwartz M, Jewelewicz R, Dyrenfurth I, Tropper P, Vande Wiele RL. The use of human menopausal and chorionic gonadotropins for induction of ovulation. Sixteen years' experience at the Sloane Hospital for Women. Am J Obstet Gynecol. 1980 Dec 1;138(7 Pt 1):801-7. doi: 10.1016/s0002-9378(16)32740-5. PMID 6778212
- [Background] Notation AD, Tagatz GE, Steffes MW. Serum 17beta-estradiol. Index of follicular maturation during gonadotropin therapy. Obstet Gynecol. 1978 Feb;51(2):204-9. PMID 622235
- [Background] Mendelson EB, Bohm-Velez M, Joseph N, Neiman HL. Gynecologic imaging: comparison of transabdominal and transvaginal sonography. Radiology. 1988 Feb;166(2):321-4. doi: 10.1148/radiology.166.2.3275976.
- [Background] Vermesh M, Kletzky OA. Follicle-stimulating hormone is the main determinant of follicular recruitment and development in ovulation induction with human menopausal gonadotropin. Am J Obstet Gynecol. 1987 Dec;157(6):1397-402. doi: 10.1016/s0002-9378(87)80231-4. PMID 3122575
- [Background] Brown JB, Evans JH, Adey FD, Taft HP, Townsend L. Factors involved in the induction of fertile ovulation with human gonadotrophins. J Obstet Gynaecol Br Commonw. 1969 Apr;76(4):289-307. doi: 10.1111/j.1471-0528.1969.tb05837.x. No abstract available. PMID 5778792
- [Background] Venturoli S, Paradisi R, Fabbri R, Magrini O, Porcu E, Flamigni C. Comparison between human urinary follicle-stimulating hormone and human menopausal gonadotropin treatment in polycystic ovary. Obstet Gynecol. 1984 Jan;63(1):6-11. PMID 6419189
- [Background] Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E. Ovarian hyperstimulation syndrome: an update review. Obstet Gynecol Surv. 1989 Jun;44(6):430-40. doi: 10.1097/00006254-198906000-00004. No abstract available. PMID 2660037